CLINICAL TRIAL: NCT05913999
Title: Prospective Evaluation of Chemotherapy-Induced Cardiotoxicity by Serial PET Myocardial Perfusion and Blood Flow Assessment - the PRECISION Trial
Brief Title: Serial PET MPI in Patients Undergoing Cancer Treatment
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rene R. Sevag Packard, MD, PhD, Assistant Professor-in-Residence, University of California, Los Angeles
Other Study IDs: IRBNet 1668650-1
Record Dates: First submitted 2023-03-17; First posted 2023-06-22 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Chemotherapeutic Toxicity; Coronary Artery Disease; Coronary Microvascular Disease
MeSH Terms: conditions — Neoplasms; Coronary Artery Disease; Microvascular Angina

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Anthracycline: Patients undergoing chemotherapy with an anthracycline-containing regimen.
- VEGF Inhibitor: Patients undergoing chemotherapy with a vascular endothelial growth factor (VEGF) inhibitor-containing regimen.
- Immune Checkpoint Inhibitor: Patients undergoing chemotherapy with an immune check point inhibitor-containing regimen.

SUMMARY:
This study aims to evaluate the effects of cardiotoxic cancer therapies on myocardial blood flow (MBF) and perfusion in a prospective sample of VA patients.

DETAILED DESCRIPTION:
Up to 60 patients who will be newly initiating chemotherapy are going to be prospectively evaluated using PET myocardial perfusion imaging (MPI) for chemotherapy-induced cardiotoxicity by quantifying MBF and perfusion. Patients will be grouped into 3 categories:

1. Patients undergoing chemotherapy with anthracycline containing regimen.
2. Patients undergoing chemotherapy with VEGF inhibitor containing regimen.
3. Patients undergoing chemotherapy with immune check point inhibitor containing regimen.

Patients will undergo PET MPI at 3 different time points:

1. Baseline PET MPI within 1 month prior to initiation of the chemotherapy regimen.
2. PET MPI at the middle of the chemotherapy regimen.
3. PET MPI within 1 month following completion of the chemotherapy regimen.

For PET MPI, the investigators will evaluate for abnormalities such as new perfusion defects, decreases in stress myocardial blood flows and decreases in myocardial flow reserves.

All study patients will also be analyzed using the following tests:

1. Echocardiogram with strain analysis within +/- 1 week of each PET MPI
2. Serology - high sensitivity troponin, cardiac C-reactive protein (CRP), brain-type natriuretic peptide (BNP), fasting lipid panel, complete metabolic panel, and complete blood count within +/- 1 week of each PET MPI study.
3. 12-lead ECG with each PET MPI study.

ELIGIBILITY:
Inclusion Criteria:

* Veterans Affairs oncology patients who will be initiating chemotherapy
* Ability to give consent

Exclusion Criteria:

* Prior chemotherapy
* Prior coronary revascularization (percutaneous coronary intervention, coronary artery bypass grafting)
* Anyone with previous invasive or CT (computed tomography) angiogram demonstrating any lesion ≥ 50% stenosis
* Known cardiomyopathy defined as rest ejection fraction < 50%
* History of heart and/or another organ transplant
* Pregnancy or breast-feeding status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cancer receiving medical care at the West Los Angeles Veterans Affairs Medical Center / Greater Los Angeles Veterans Affairs Healthcare System.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
PET myocardial perfusion imaging (MPI). | Baseline (within 1 month prior to the initiation of cancer treatment), during cancer treatment (estimated at 1-6 months), and within 1 month post-cancer treatment completion (approximately 2-9 months)
  Change from baseline in number of patients with perfusion defects measured as % total perfusion deficit (TPD) of the left ventricular myocardium by PET
PET myocardial blood flow (MBF) measurement. | Baseline (within 1 month prior to the initiation of cancer treatment), during cancer treatment (estimated at 1-6 months), and within 1 month post-cancer treatment completion (approximately 2-9 months)
  Change from baseline in number of patients with myocardial blood flow abnormalities measured as stress myocardial blood flow (SMBF) values < 2 mL/min/g of left ventricular myocardium by PET

SECONDARY OUTCOMES:
Transthoracic echocardiography (TTE) global left ventricular systolic function. | Baseline (within 1 month prior to the initiation of cancer treatment), during cancer treatment (estimated at 1-6 months), and within 1 month post-cancer treatment completion (approximately 2-9 months)
  Change from baseline in number of patients with global systolic dysfunction measured as % left ventricular ejection fraction by TTE.
Transthoracic echocardiography (TTE) focal left ventricular systolic function. | Baseline (within 1 month prior to the initiation of cancer treatment), during cancer treatment (estimated at 1-6 months), and within 1 month post-cancer treatment completion (approximately 2-9 months)
  Change from baseline in number of patients with focal systolic dysfunction measured as % left ventricular global longitudinal strain by TTE.
Transthoracic echocardiography (TTE) focal left atrial systolic function. | Baseline (within 1 month prior to the initiation of cancer treatment), during cancer treatment (estimated at 1-6 months), and within 1 month post-cancer treatment completion (approximately 2-9 months)
  Change from baseline in number of patients with focal systolic dysfunction measured as % left atrial strain by TTE.
Electrocardiogram (ECG) findings. | Baseline (within 1 month prior to the initiation of cancer treatment), during cancer treatment (estimated at 1-6 months), and within 1 month post-cancer treatment completion (approximately 2-9 months)
  Change from baseline in number of patients with any of the following ECG changes:
  * new T-wave inversions
  * new ST-segment deviations >/= 1mm
  * new left bundle branch block
Metabolic or cardiac function abnormalities as determined by blood work findings | Baseline (within 1 month prior to the initiation of cancer treatment), during cancer treatment (estimated at 1-6 months), and within 1 month post-cancer treatment completion (approximately 2-9 months)
  Change from baseline in number of patients with changes in the values of serological tests indicative of metabolic or cardiac function abnormalities including one or more of the following:
  * high sensitivity troponin (ng/L)
  * cardiac C-reactive protein (mg/L)
  * brain-type natriuretic peptide (pg/mL)
  * fasting lipid panel: total cholesterol (mg/dL), low-density lipoprotein cholesterol (mg/dL), high-density lipoprotein cholesterol (mg/dL), triglycerides (mg/dL)
  * complete metabolic panel: total protein (g/dL), albumin (g/dL), total bilirubin (mg/dL), direct bilirubin (mg/dL), aspartate aminotransferase (IU/L), alanine transaminase (IU/L), alkaline phosphatase (IU/L), sodium (mmol/L), potassium (mmol/L), chloride (mmol/L), bicarbonate (mmol/L), blood urea nitrogen (mg/dL), creatinine (mg/dL), glucose (mg/dL)
  * complete blood count: white blood cell count (k/uL), hemoglobin (g/dL), hematocrit (%), platelet (k/uL)

CONTACTS AND LOCATIONS:
Overall Officials: Rene Packard, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- West Los Angeles VA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Herrmann J, Yang EH, Iliescu CA, Cilingiroglu M, Charitakis K, Hakeem A, Toutouzas K, Leesar MA, Grines CL, Marmagkiolis K. Vascular Toxicities of Cancer Therapies: The Old and the New--An Evolving Avenue. Circulation. 2016 Mar 29;133(13):1272-89. doi: 10.1161/CIRCULATIONAHA.115.018347. PMID 27022039
- [Background] Chang HM, Moudgil R, Scarabelli T, Okwuosa TM, Yeh ETH. Cardiovascular Complications of Cancer Therapy: Best Practices in Diagnosis, Prevention, and Management: Part 1. J Am Coll Cardiol. 2017 Nov 14;70(20):2536-2551. doi: 10.1016/j.jacc.2017.09.1096. PMID 29145954
- [Background] Hader SN, Zinkevich N, Norwood Toro LE, Kriegel AJ, Kong A, Freed JK, Gutterman DD, Beyer AM. Detrimental effects of chemotherapy on human coronary microvascular function. Am J Physiol Heart Circ Physiol. 2019 Oct 1;317(4):H705-H710. doi: 10.1152/ajpheart.00370.2019. Epub 2019 Aug 9. PMID 31397169
- [Background] Yeh ET, Bickford CL. Cardiovascular complications of cancer therapy: incidence, pathogenesis, diagnosis, and management. J Am Coll Cardiol. 2009 Jun 16;53(24):2231-47. doi: 10.1016/j.jacc.2009.02.050. PMID 19520246
- [Background] Murthy VL, Bateman TM, Beanlands RS, Berman DS, Borges-Neto S, Chareonthaitawee P, Cerqueira MD, deKemp RA, DePuey EG, Dilsizian V, Dorbala S, Ficaro EP, Garcia EV, Gewirtz H, Heller GV, Lewin HC, Malhotra S, Mann A, Ruddy TD, Schindler TH, Schwartz RG, Slomka PJ, Soman P, Di Carli MF; SNMMI Cardiovascular Council Board of Directors; ASNC Board of Directors. Clinical Quantification of Myocardial Blood Flow Using PET: Joint Position Paper of the SNMMI Cardiovascular Council and the ASNC. J Nucl Med. 2018 Feb;59(2):273-293. doi: 10.2967/jnumed.117.201368. Epub 2017 Dec 14. No abstract available. PMID 29242396
- [Background] Murthy VL, Naya M, Foster CR, Hainer J, Gaber M, Di Carli G, Blankstein R, Dorbala S, Sitek A, Pencina MJ, Di Carli MF. Improved cardiac risk assessment with noninvasive measures of coronary flow reserve. Circulation. 2011 Nov 15;124(20):2215-24. doi: 10.1161/CIRCULATIONAHA.111.050427. Epub 2011 Oct 17. PMID 22007073
- [Background] Ziadi MC, Dekemp RA, Williams KA, Guo A, Chow BJ, Renaud JM, Ruddy TD, Sarveswaran N, Tee RE, Beanlands RS. Impaired myocardial flow reserve on rubidium-82 positron emission tomography imaging predicts adverse outcomes in patients assessed for myocardial ischemia. J Am Coll Cardiol. 2011 Aug 9;58(7):740-8. doi: 10.1016/j.jacc.2011.01.065. PMID 21816311